CLINICAL TRIAL: NCT06765681
Title: SepThrom: Exploring the Relationship Between Sepsis, VTE and DIC in RWD.
Brief Title: An Observational Study in the United States to Learn How Venous Thromboembolism, Disseminated Intravascular Coagulation, and Sepsis Are Related
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22892
Record Dates: First submitted 2024-12-16; First posted 2025-01-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Venous Thromboembolism; Disseminated Intravascular Coagulation
MeSH Terms: conditions — Sepsis; Venous Thromboembolism; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diagnosed DIC: Patients with ICD10 (International Classification of Diseases) code for DIC
  Interventions: Other: Diagnosis of both VTE and sepsis
- Undiagnosed DIC: Patients with SIC (Sepsis Induced Coagulopathy) score of >/= 4
  Interventions: Other: Diagnosis of both VTE and sepsis
- No DIC: Patients with no DIC within the same hospital stay
  Interventions: Other: Diagnosis of both VTE and sepsis

INTERVENTIONS:
Other: Diagnosis of both VTE and sepsis — Both diagnoses need to present during ICU stay for case inclusion into this retrospective study

SUMMARY:
This is an observational study in which data already collected from people with venous thromboembolism (VTE) due to sepsis (blood poisoning) are studied. These people were hospitalized in an intensive care unit (ICU) and may or may not have had disseminated intravascular coagulation (DIC).

In this observational study, only observations are made without participants receiving any advice or changes to their healthcare.

VTE is a condition that occurs when blood clots form in the veins, which can be dangerous. DIC is a serious blood disorder that can cause clots throughout the body, blocking blood flow. People who have sepsis are at a higher risk of developing both VTE and DIC. Researchers wanted to know if people who have sepsis developed DIC before developing VTE.

To prevent VTE in people with sepsis, it is important to know how severe the sepsis is, how it progresses, and whether DIC is also present or not.

In this study, researchers will assess patient data from a medical database in the United States (US).

The main purpose of this study is to learn if there is a relationship between sepsis, DIC, and VTE.

To do this, researchers will divide the participants with VTE due to sepsis into three groups as follows:

* participants who were diagnosed with DIC based on the extent of blood clotting
* participants who likely had DIC but it was not diagnosed
* participants who did not develop DIC during the same hospital visit

The researchers will collect the following information:

* the number of participants who had VTE due to sepsis also had DIC
* the change in participants' laboratory results and vital signs, such as heart rate and blood pressure, from the time their sepsis was diagnosed to the time their VTE and DIC were diagnosed

The researchers will study the data collected between January 2007 and December 2021.

The data will come from the participants' information stored in a database called the Optum VTE EHR which collects patient medical data from hospitals across the US.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* admitted to an ICU with the diagnosis of VTE and sepsis during the same hospital ICU admission

Exclusion Criteria:

* less than 18 yrs old
* less than 365 days data available prior to index VTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All inpatients admitted to an ICU with the diagnosis of VTE and sepsis during the same hospital ICU admission, within the Optum VTE EHR dataset from 1 January 2007 to 31 December 2021
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of diagnosed DIC among hospitalized people with sepsis-associated VTE | Retrospective analysis of 15 year dataset
Proportion of undiagnosed DIC among hospitalized people with sepsis-associated VTE | Retrospective analysis of 15 year dataset
  Based on trajectory of laboratory and vital sign data from the time of sepsis ICD10 coding to the time of VTE coding and to the time of DIC coding

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.